CLINICAL TRIAL: NCT06382584
Title: Impact of Treatment With Direct Oral Anticoagulants (Anti Xa) on the Management and Outcome of Patients With Fractures of the Upper End of the Femur: Retrospective Analysis of Nimes University Hospital Database
Brief Title: Impact of Treatment With Oral Anticoagulants of Patients With Fractures of the Upper End of the Femur
Acronym: ANTI_XA AOD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB_23.09.01
Record Dates: First submitted 2023-12-06; First posted 2024-04-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Direct Oral Anticoagulants (DOACs); Femoral Fractures; Surgery
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti XA: adults treated with direct oral factor Xa inhibitors undergoing Femoral head fracture surgery
  Interventions: Procedure: Femoral fracture surgery

INTERVENTIONS:
Procedure: Femoral fracture surgery — Hip fracture surgery

SUMMARY:
In 2023, oral anticoagulant treatments (anti Xa: apixaban , rivaroxaban, etc.) are tending to replace anti vitamin K treatments in many medical indications. Their prescription is increasing rapidly in the elderly.

In this context, the Nimes University Hospital receives a large number of elderly patients who have suffered a fracture of the end of the femur requiring surgery and who are taking anti Xa drugs.To avoid massive intra- and post-operative haemorrhage, surgical management is postponed because of the need to suspend the treatment, allowing a return to near-normal biological haemostasis within a few days. No consensus has been reached on the withdrawal period required to authorise surgery, as the elimination kinetics of the drug are altered in this context (elderly patients, dehydration, hypovolaemia, impaired renal function). A plasma assay (threshold of <30 to 60 ng/mL) has been proposed without any real justification. This waiting period exposes the elderly to excess mortality. Reversing these treatments by adding coagulation factors would be an attractive alternative, as it would allow surgery to be performed earlier, but this would expose patients to an increased thrombotic risk.

Before considering a prospective randomised study (early vs delayed surgery on AOD), we wish to retrospectively analyse data on patients admitted to the Nimes University Hospital on anti Xa and operated on for fracture of the upper end of the femur between 1 January 2022 and 1 June 2023

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 65 years
* Emergency admission for isolated fracture of the upper end of the femur
* Requires osteosynthesis surgery
* Hospitalized in geriatric perioperative unit, chu Nimes (UPOG)
* On anti Xa therapy prior to hospitalisation

Exclusion Criteria:

* Patients under court order or not affiliated to a social security scheme
* Outpatient surgery
* Multiple fractures and/or other associated surgery
* Not admitted to UPOG
* No surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly Patients treated with direct oral factor Xa inhibitors requiring osteosynthesis surgery for isolated fracture of the upper end of the femur recorded in Nimes University Hospital database between January 1, 2022 and June 1, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | Day 0 to Day 28
  hospital mortality within 28 days of the date of hospital admission for femoral head fracture

SECONDARY OUTCOMES:
Duration of the surgery | During surgery
  Time required for surgery
Transfusion | Day 0 to Day 28
  Need for a transfusion
Postoperative comorbidities | Day 0 to Day 28
  postoperative comorbidities during surgery and until day 28
Hospital stay | Day 0 to Day 28
  length of hospital stay
Anti Xa assay | Day 0 to Day 28
  anti Xa assay during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, Principal Investigator — CHU NIMES
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gricourt Y, Perin M, Basseres N, Geronimi L, Lefrant JY, Mezzarobba M, Chea M, Gris JC, Cuvillon P. Impact of direct oral anticoagulant treatment on management and outcomes of patients with hip fractures by monitoring assays. A population-based study of a cohort from the Geriatric Perioperative Unit. Anaesth Crit Care Pain Med. 2026 Jan;45(1):101616. doi: 10.1016/j.accpm.2025.101616. Epub 2025 Oct 4. PMID 41052671